CLINICAL TRIAL: NCT06929598
Title: The Efficacy of Adjunctive Shiatsu Therapy for Non-Inflammatory Chronic Pain in Pediatric Patients: A Single-Arm Prospective Trial
Brief Title: Shiatsu for Chronic Non-Inflammatory Pain in Children and Adolescents
Acronym: ShiQoL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: Tel Aviv Sourasky Medical Center, Tel Aviv, Israel (Unknown); Dana-Dwek Children's Hospital (Unknown)
Responsible Party: Principal Investigator, Eyal Cohen-Sela, Medical Doctor, Tel Aviv University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0661-2222
Record Dates: First submitted 2025-04-01; First posted 2025-04-16 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain; Chronic Pain Syndrome; Chronic Pain and Comorbid Emotional Problems; Chronic Pain, Psychogenic; Chronic Pain, Widespread; Fibromyalgia; Fibromyalgia Syndrome; Functional Pain
Keywords: Shiatsu; Complementary and Integrative Medicine; Pediatric Chronic Pain; Non-inflammatory Pain; Quality of Life; PedsQL; Adolescent Pain; Manual Therapy; Mind-Body Therapy; Pediatric Rheumatology; Integrative Medicine; Functional Pain; Pain Management
MeSH Terms: conditions — Chronic Pain; Fibromyalgia; Agnosia | interventions — Hydrotherapy

STUDY DESIGN:
Intervention Model Description: This is a single-arm, prospective study evaluating the effects of adjunctive Shiatsu therapy on quality of life in children and adolescents with non-inflammatory chronic pain. All participants receive the same intervention without a comparison or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Shiatsu Therapy Group (Experimental): Participants will receive 30-minute Shiatsu therapy sessions once a week for 6 weeks, in addition to their usual pain management. The goal is to assess whether Shiatsu improves quality of life in children and adolescents with non-inflammatory chronic pain.
  Interventions: Behavioral: Shiatsu Therapy

INTERVENTIONS:
Behavioral: Shiatsu Therapy — Participants will receive one 30-minute session of Shiatsu therapy per week for 6 weeks. Therapy will be provided by trained Shiatsu practitioners under a standardized protocol developed for this study.

SUMMARY:
The goal of this clinical trial is to learn if adding Shiatsu therapy to standard treatment can improve quality of life in children and adolescents with chronic pain that is not caused by inflammation. The main question it aims to answer is: Does Shiatsu therapy help improve the quality of life in children with long-lasting pain?

All participants will continue their regular treatment and will also:

* Receive a 30-minute Shiatsu session once a week for six weeks
* Complete questionnaires about their quality of life and family impact before, during, and after the treatment period

The study includes about 40 participants between the ages of 10 and 18, who are already being followed at the pediatric pain and rheumatology clinics at Tel Aviv Sourasky Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 10-18 years
* Diagnosed with non-inflammatory chronic pain syndromes
* Actively followed by the Pediatric Rheumatology and/or Pediatric Pain Clinics at Tel Aviv Sourasky Medical Center (at least twice a year)
* Informed consent signed by at least one legal guardian (or both guardians in cases of separated parents)
* If participant is 16 years or older, they must also sign the informed consent

Exclusion Criteria:

* Informed consent cannot be obtained from the participant or their legal guardians
* Legal guardians unable to provide informed consent
* Patients with severe conditions (e.g., bone metastasis)
* Patients unable to participate in Shiatsu therapy sessions
* Participation in Shiatsu therapy within 6 months prior to study enrollment
* Participant or legal guardian refuses participation

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pediatric Quality of Life Inventory Version 4.0 (PedsQL 4.0) Generic Core Scale Total Score | Baseline (Day 0), Week 3 (after the 3rd Shiatsu session), Week 6 (after the 6th Shiatsu session, end of intervention), and Week 18 (3 months post-intervention)
  The PedsQL 4.0 Generic Core Scale is a validated questionnaire that measures health-related quality of life in children and adolescents. Participants will complete the age-appropriate version of the PedsQL. It includes 23 items across four subscales: physical, emotional, social, and school functioning. Responses are reverse-scored and transformed to a 0-100 scale. Higher scores indicate better quality of life. The change in total score from baseline to follow-up time points will be assessed.

SECONDARY OUTCOMES:
Change in Pediatric Quality of Life Inventory Family Impact Module (PedsQL FIM) Total Score | Baseline (Day 0), Week 3 (after the 3rd Shiatsu session), Week 6 (after the 6th Shiatsu session, end of intervention), and Week 18 (3 months post-intervention)
  The Pediatric Quality of Life Inventory Family Impact Module (PedsQL FIM) is a validated caregiver-reported questionnaire that assesses the impact of a child's health condition on family functioning. It includes 36 items covering physical, emotional, social, and cognitive functioning, communication, worry, daily activities, and family relationships. Responses are reverse-scored and transformed to a 0-100 scale. Higher scores indicate better family functioning and less caregiver burden. The change in total score from baseline to follow-up time points will be assessed.
Change in Pain Intensity (Numerical Rating Scale, NRS) | Baseline (Day 0), Week 3 (after the 3rd Shiatsu session), Week 6 (after the 6th Shiatsu session, end of intervention), and Week 18 (3 months post-intervention)
  Pain intensity will be self-reported using the Numerical Rating Scale (NRS), a validated 11-point scale ranging from 0 to 10, where 0 means "no pain" and 10 means "worst possible pain." Participants will rate their pain at each time point. The change in score from baseline to follow-up time points will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Merav Heshin-Bekenstein, MD, Principal Investigator — Dana Dwek Children's Hospital, Tel Aviv Medical Center, Tel Aviv University, Tel Aviv, Israel
Locations (2):
- Israel (2):
  - Tel Aviv Univrsity, Tel Aviv, Tel Aviv
  - Dana-Dwek Children's Hospital, Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: Undecided
The research team has not yet finalized a plan for sharing individual participant data (IPD). Data sharing options will be considered in accordance with institutional board review, policies, ethical guidelines in our institution, ethical guidelines for pediatric research, and data privacy regulations.